CLINICAL TRIAL: NCT06298929
Title: Medial Rectus Muscle Fenestration Versus Medial Rectus Recession for Partially Accommodative Esotropia
Brief Title: Medial Rectus Fenestration vs Recession for PAET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Ameera Gamal Abdelhameed, assistant professor of ophthalmology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR427/11/23
Record Dates: First submitted 2024-02-25; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Partially Accommodative Esotropia
Keywords: esotropia; accommodative; hyperopia; recession; fenestration
MeSH Terms: conditions — Esotropia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): patients with PAET who will receive unilateral or bilateral MR fenestration
  Interventions: Procedure: medial rectus fenestration
- Group 2 (Active Comparator): patients with PAET who will receive unilateral or bilateral MR recession
  Interventions: Procedure: medial rectus recession

INTERVENTIONS:
Procedure: medial rectus fenestration — Fenestration technique involves making two splitting incisions by blunt dissection parallel to the muscle fibers on the superior and inferior borders of the muscle, leaving 1 mm of muscle fibers on each edge. The rectangular wide central part is excised from the insertion and between the two splitting incisions to a point back 5-8 mm depending on the angle of the esotropia.
  Arms: Group 1
Procedure: medial rectus recession — recession is one of the gold standard weakening procedures that involves disinsertion of the muscle and re-suturing to the sclera at a more posterior location to decrease its contractile power.
  Arms: Group 2

SUMMARY:
This prospective comparative study aims to compare medial rectus (MR) muscle fenestration and recession in patients with partially accommodative esotropia (PAET). The main question it aims to answer is whether MR fenestration is equally effective as MR recession for PAET.

All patients will receive complete ophthalmic and orthoptic assessment. Patients will be randomly allocated using a random table to one of two groups; Group 1 will receive conventional MR recession, and Group 2 will receive MR fenestration.

DETAILED DESCRIPTION:
Inclusion criteria The study will include patients with accommodative esotropia if the residual distance deviation with full cycloplegic correction is > 15PD.

Exclusion criteria:

1. Patients with convergence excess esotropia, defined as a near deviation with glasses exceeding that for distance by 15 PD or more.
2. Patients with paralytic or restrictive strabismus.
3. Patients with previous strabismus surgery
4. Patients with neurologic, ocular, or developmental disorders or follow-up less than 6 months

All patients will receive complete ophthalmic and orthoptic assessment including:

i) A full ophthalmological assessment including history taking, measurement of uncorrected and best-corrected visual acuity, cycloplegic refraction, anterior segment examination, as well as a dilated fundus examination.

ii) Measurement of the deviation at distance (6 m) and near (33 cm). iii) Assessment of ductions and versions in all cardinal directions of gaze

Patients will be randomly allocated using a random table to one of two groups:

1. Group 1: Unilateral or bilateral conventional MR recession. Augmented formula will be used to decide the Surgical dosage using the standard tables (3)
2. Group 2: unilateral or bilateral MR fenestration All surgeries will be performed by one experienced surgeon (H.SH)

ELIGIBILITY:
Inclusion Criteria:

* patients with accommodative esotropia if the residual distance deviation with full cycloplegic correction is > 15PD.

Exclusion Criteria:

1. convergence excess esotropia.
2. paralytic or restrictive strabismus.
3. previous strabismus surgery
4. neurologic, ocular, or developmental disorders or follow-up less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Ocular alignment (measured in prism diopters) | 6 months postoperative
  The distance and near angles of deviation, with and without glasses, and the angle disparity

SECONDARY OUTCOMES:
ocular motility | 6 months postoperative
  ductions of both eyes (graded on a scale of nine points from -4 to +4)

CONTACTS AND LOCATIONS:
Overall Officials: Ameera G Abdelhameed, MD, Principal Investigator — Assistant professor of ophthalmology
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No